CLINICAL TRIAL: NCT06049017
Title: A Phase 2b Multicenter, Randomized, Placebo- Controlled, Dose-Ranging Study to Evaluate the Efficacy and Safety of JNJ-77242113 for the Treatment of Moderately to Severely Active Ulcerative Colitis
Brief Title: A Study of JNJ-77242113 in Participants With Moderately to Severely Active Ulcerative Colitis
Acronym: ANTHEM-UC
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 77242113UCO2001; 77242113UCO2001 (Other: Janssen Research & Development, LLC); 2023-504673-20-00 (Registry Identifier: EUCT number)
Record Dates: First submitted 2023-09-15; First posted 2023-09-21 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Colitis, Ulcerative
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Group 1: JNJ-77242113 Dose-1 (Experimental): Participants will receive JNJ-77242113 Dose-1 tablets orally from Week 0 through Week 28. Participants who complete the Week 28 assessments and have achieved clinical response at Week 28 and who, in the opinion of the investigator, will continue to benefit from treatment with study intervention will continue in the 48-week long term extension (LTE) period and receive the same treatment up to Week 76.
  Interventions: Drug: JNJ-77242113
- Group 2: JNJ-77242113 Dose-2 (Experimental): Participants will receive JNJ-77242113 Dose-2 tablets orally from Week 0 through Week 28. Participants who complete the Week 28 assessments and have achieved clinical response at Week 28 and who, in the opinion of the investigator, will continue to benefit from treatment with study intervention will continue in the 48-week LTE period and receive the same treatment up to Week 76.
  Interventions: Drug: JNJ-77242113
- Group 3: JNJ-77242113 Dose-3 (Experimental): Participants will receive JNJ-77242113 Dose-3 tablets orally from Week 0 through Week 28. Participants who complete the Week 28 assessments and have achieved clinical response at Week 28 and who, in the opinion of the investigator, will continue to benefit from treatment with study intervention will continue in the 48-week LTE period and receive the same treatment up to Week 76.
  Interventions: Drug: JNJ-77242113
- Group 4: Placebo (Experimental): Participants will receive placebo tablets orally from Week 0 through Week 28. Placebo-treated participants who meet the criteria of inadequate response at Week 16, will receive JNJ-77242113 Dose-3 tablet orally through Week 28. Participants who complete the Week 28 assessments and have achieved clinical response at Week 28 and who, in the opinion of the investigator, will continue to benefit from treatment with study intervention, will continue in the 48-week LTE period and receive the same treatment up to Week 76.
  Interventions: Drug: JNJ-77242113; Drug: Placebo

INTERVENTIONS:
Drug: JNJ-77242113 — JNJ-77242113 tablet will be administered orally.
Drug: Placebo — Placebo tablet will be administered orally.
  Arms: Group 4: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of JNJ-77242113 compared with placebo in participants with moderately to severely active ulcerative colitis.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form 18 years of age or older
* Documented diagnosis of ulcerative colitis (UC) of at least 12 weeks prior to screening
* Moderately to severely active UC as per the modified Mayo score
* Demonstrated inadequate response to or intolerance of conventional therapy and/or advanced therapy as defined in the protocol

Exclusion Criteria:

* Participants with current or prior diagnosis of fulminant colitis and/or toxic megacolon
* UC limited to rectum only or to less than (<) 15 centimeters (cm) of colon
* Presence of a stoma
* Presence or history of fistula
* History of extensive colonic resection (example, <30 cm of colon remaining)
* Diagnosis of indeterminate colitis, microscopic colitis, ischemic colitis, Crohn's colitis or clinical findings suggestive of Crohn's disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 252 (Actual)
Dates: Start 2023-10-09 (Actual); Primary Completion 2024-09-26 (Actual); Study Completion 2026-01-16 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants with Clinical Response at Week 12 | Week 12
  Clinical response is defined as decrease from baseline in the modified Mayo score by greater than or equal to (>=) 30 percent (%) and >=2 points, with either a >=1-point decrease from baseline in the rectal bleeding subscore or a rectal bleeding subscore of 0 or 1.

SECONDARY OUTCOMES:
Percentage of Participants with Clinical Remission at Week 12 | Week 12
  Clinical remission is defined as stool frequency subscore of 0 or 1, where the stool frequency subscore has not increased from baseline, a rectal bleeding subscore of 0, and an endoscopy subscore of 0 or 1.
Percentage of Participants with Symptomatic Remission at Week 12 | Week 12
  Symptomatic remission is defined as stool frequency subscore of 0 or 1, where the stool frequency subscore has not increased from baseline, and a rectal bleeding subscore of 0.
Percentage of Participants with Endoscopic Improvement at Week 12 | Week 12
  Endoscopic improvement is defined as an endoscopy subscore of 0 or 1.
Percentage of Participants with Histologic-endoscopic Mucosal Improvement at Week 12 | Week 12
  Histologic-endoscopic mucosal improvement is defined as a combination of histologic remission and endoscopic improvement. Histologic remission and endoscopic improvement are based on the histologic grading and the Mayo endoscopy subscore.
Percentage of Participants with Adverse Events (AE) and Serious Adverse Evets (SAEs) | Up to Week 76
  An AE is any untoward medical occurrence in a clinical study participant administered a pharmaceutical (investigational or non-investigational) product. An AE does not necessarily have a causal relationship with the intervention. A SAE is any untoward medical occurrence that at any dose: results in death; is life-threatening; requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity; is a congenital anomaly/birth defect; is a suspected transmission of any infectious agent via a medicinal product; is medically important.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (176):
- United States (32):
  - Clinnova Research, Anaheim, California
  - Hoag Memorial Hospital, Newport Beach, California
  - Medical Associates Research Group, Inc., San Diego, California
  - Peak Gastroenterology Associates, Colorado Springs, Colorado
  - I.H.S. Health. LLC, Kissimmee, Florida
  - Endoscopic Research Inc, Orlando, Florida
  - GCP Clinical Research, Tampa, Florida
  - Atlanta Gastroenterology Associates, Atlanta, Georgia
  - Gastroenterology of Southern Indiana, New Albany, Indiana
  - Cotton O'Neil Digestive Health Center, Topeka, Kansas
  - Ochsner Medical Center, Jefferson, Louisiana
  - Tandem Clinical Research, Marrero, Louisiana
  - Mercy Medical Center, Baltimore, Maryland
  - Mayo Clinic Rochester, Rochester, Minnesota
  - New York Gastroenterology Associates, New York, New York
  - DiGiovanna Institute for Medical Education & Research, North Massapequa, New York
  - University North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Atrium Health, Charlotte, North Carolina
  - Charlotte Gastroenterology and Hepatology, PLLC, Charlotte, North Carolina
  - Northshore Gastroenterology Research, LLC, Westlake, Ohio
  - Digestive Disease Specialists Inc, Oklahoma City, Oklahoma
  - Gastroenterology Associates P.A., Greenville, South Carolina
  - DHAT Research Institute, Garland, Texas
  - Amel Med LLC Research, Georgetown, Texas
  - Accurate Clinical Research, Inc., Humble, Texas
  - Caprock Gastro Research, Lubbock, Texas
  - Southern Star Research Institute, LLC, San Antonio, Texas
  - Tyler Research Institute, LLC, Tyler, Texas
  - Care Access Research, Ogden, Ogden, Utah
  - Gastroenterology Associates of Tidewater, Chesapeake, Virginia
  - Washington Gastroenterology, PLLC, Bellevue, Washington
  - Washington Gastroenterology, PLLC, Tacoma, Washington
- Argentina (5):
  - Cer Instituto Medico, Buenos Aires
  - CIPREC, Buenos Aires
  - Gedyt - Consultorios Gastroenterologia, Buenos Aires
  - Hospital Provincial del Centenario, Rosario
  - Sanatorio 9 de Julio, San Miguel de Tucumán
- Australia (4):
  - Sunshine Coast University Hospital, Birtinya
  - Blacktown Hospital, Blacktown
  - Concord Repatriation General Hospital, Concord
  - Wollongong Private Hospital, Wollongong
- Belgium (6):
  - CHU Saint-Pierre, Brussels
  - AZ Sint-Lucas, Ghent
  - Ghent University Hospital, Ghent
  - Universitair Ziekenhuis Leuven, Leuven
  - Centre Hospitalier Universitaire de Liege Domaine Universitaire du Sart Tilman, Liège
  - Vitaz, Sint-Niklaas
- Brazil (8):
  - UNESP - Faculdade de Medicina da Universidade Estadual Paulista - Campus Botucatu, Botucatu
  - L2IP Instituto de Pesquisas Clinicas, Brasília
  - CDC - Centro Digestivo de Curitiba, Curitiba
  - Hospital de Clinicas de Porto Alegre - Hospital de Clinicas, Porto Alegre
  - Pesquisare Saude, Santo André
  - BR TRIALS Ensaios Clinicos e Consultoria Ltda, São Paulo
  - Instituto D Or de Pesquisa e Ensino, São Paulo
  - INTEGRAL Pesquisa e Ensino, Votuporanga
- Canada (5):
  - Gastroenterology and Internal Medicine Research Institute (GIRI), Edmonton, Alberta
  - Barrie GI Associates, Barrie, Ontario
  - London Health Sciences Centre, London, Ontario
  - ABP Research Services Corp., Oakville, Ontario
  - Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec
- China (12):
  - The second Xiangya Hospital of Central South University, Changsha
  - Chongqing General Hospital, Chongqing
  - The First Affiliated Hospital Sun Yat sen University, Guangzhou
  - The Sixth Affiliated Hospital Sun Yat sen University, Guangzhou
  - Sir Run Run Shaw Hospital Zhejiang University School of Medicine, Hangzhou
  - Qilu Hospital of Shandong University, Jinan
  - Lanzhou University Second Hospital, Lanzhou
  - Nanjing Drum Tower Hospital, Nanjing
  - Shengjing Hospital Of China Medical University, Shenyang
  - Union Hospital Tongji Medical College of Huazhong University of Science and Technology, Wuhan
  - Wuxi People s Hospital, Wuxi
  - The Second Affiliated Hospital of Air Force Medical University - Tangdu Hospital, Xi'an
- Czechia (5):
  - Nemocnice Ceske Budejovice, České Budějovice
  - Gastroenterologie, s.r.o., Hradec Kralove, Hradec Kralova
  - Hepato-gastroenterologie HK, s.r.o., Hradec Králové
  - ISCARE a.s., Prague
  - Nemocnice Slany, Slaný
- France (11):
  - CHRU Besancon Hopital Jean Minjoz, Besançon
  - APHP - Hopital Henri Mondor, Créteil
  - CHRU de Lille Hopital Claude Huriez, Lille
  - Clinique Ambroise Pare, Neuilly-sur-Seine
  - CHU de Nice Hopital de l Archet, Nice
  - CHU Nimes Hopital Caremeau, Nîmes
  - APHP - Hopital Bichat - Claude Bernard, Paris
  - Hospices Civils de Lyon CHU Lyon Sud, Pierre-Bénite
  - CHU Saint Etienne Hopital Nord, Saint-Priest-en-Jarez
  - CHU Toulouse - Hopital de Rangueil, Toulouse
  - CHU de Nancy_ Hopital Brabois, Vandœuvre-lès-Nancy
- Germany (8):
  - Klinikum Augsburg, Augsburg
  - Krankenhaus Waldfriede Mitte, Berlin
  - Universitaetsklinikum Carl Gustav Carus TU Dresden, Dresden
  - Medizinische Hochschule Hannover, Hanover
  - Universitatsklinikum Schleswig Holstein Kiel, Kiel
  - Eugastro GmbH, Leipzig
  - Staedtisches Klinikum Lueneburg, Lüneburg
  - Gastroenterologische Gemeinschaftspraxis Minden, Minden
- Hungary (5):
  - Semmelweis Egyetem, Budapest
  - Pannónia Magánorvosi Centrum Kft, Budapest
  - Vasutegeszsegugyi Nonprofit Kozhasznu Kft, Debrecen
  - Debreceni Egyetem Gasztroenterologiai Klinika, Debrecen
  - Clinexpert Kft, Gyöngyös
- India (4):
  - S. R. Kalla Memorial General Hospital, Jaipur
  - Midas Hospital, Nagpur
  - Govind Ballabh Pant Hospital, New Delhi
  - SIDS Hospital & Research Centre, Surat
- Italy (7):
  - Fondazione IRCCS Ca Granda Ospedale Policlinico Di Milano, Milan
  - Ospedale San Raffaele di Milano, Milan
  - Ospedale Sacro Cuore Don Calabria, Negrar
  - Azienda Ospedaliera San Camillo - Roma, Roma
  - Fondazione Policlinico Universitario A Gemelli IRCCS, Roma
  - Istituto Clinico Humanitas, Rozzano
  - Casa Sollievo Della Sofferenza IRCCS, San Giovanni Rotondo
- Japan (14):
  - Sai Gastroenterology Proctology, Fujiidera-shi
  - Hamamatsu University Hospital, Hamamatsu
  - Kagoshima IBD Gastroenterology Clinic, Kagoshima
  - Tsujinaka Hospital Kashiwanoha, Kashiwa
  - Aoyama Naika Clinic, Kobe
  - Kinshukai Infusion Clinic, Osaka
  - Japanese Red Cross Osaka Hospital, Osaka
  - Toho University Sakura Medical Center, Sakura
  - Sapporo Tokushukai Hospital, Sapporo
  - Sapporo Higashi Tokushukai Hospital, Sapporo
  - National Hospital Organization Shizuoka Medical Center, Shimizu
  - Tokyo Metropolitan Bokutoh Hospital, Sumida Ku
  - Mie University Hospital, Tsu
  - Yokohama City University Medical Center, Yokohama
- Malaysia (3):
  - Hospital Sultanah Aminah, Johor Bahru
  - Sultan Idris Shah Hospital, Kajang
  - University Malaya Medical Centre, Kuala Lumpur
- Poland (12):
  - Centrum Medyczne Medis ManerMed Sp Z O O, Bydgoszcz
  - Centrum Medyczne Lukamed Spolka z Ograniczona Odpowiedzialnoscia, Chojnice
  - Centrum Medyczne Plejady, Krakow
  - Centrum Medyczne Medyk, Rzeszów
  - Sonomed Sp. z o.o., Szczecin
  - GASTROMED Sp. z o.o., Torun
  - Centralny Szpital Kliniczny Mswia, Warsaw
  - Bodyclinic Sp. z o.o. sp. k, Warsaw
  - Medical Network Spolka z o.o. WIP Warsaw IBD Point Profesor Kierkus, Warsaw
  - Centrum Medyczne Oporow, Wroclaw
  - Melita Medical Sp. z o.o., Wroclaw
  - EMC Instytut Medyczny SA, Wroclaw
- Romania (4):
  - Spital Memorial, Bucharest
  - S C Delta Health Care S R L, Bucharest
  - Digenio - Centrul Medical de Gastroenterologie, Hepatologie si Endoscopie Digestiva, Cluj-Napoca
  - Centrul Medical Valahia, Ploieşti
- South Korea (7):
  - Inje University Haeundae Paik Hospital, Busan
  - Yeungnam University Hospital, Daegu
  - Seoul National University Hospital, Seoul
  - Kangbuk Samsung Hospital, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic university of Korea, St. Vincent's Hospital, Suwon
- Spain (11):
  - Hosp. Univ. Fundacion Alcorcon, Alcorcón
  - Hosp. Arquitecto Marcide, Ferrol
  - Hosp. de Cabuenes, Gijón
  - Hosp. Univ. La Paz, Madrid
  - Hosp. Univ. Pta. de Hierro Majadahonda, Majadahonda
  - Hosp. Clinico Univ. de Santiago, Santiago de Compostela
  - Hosp. Virgen Macarena, Seville
  - Hosp. Ntra. Sra. de Valme, Seville
  - Hosp. Clinico Univ. de Valencia, Valencia
  - Hosp. Univ. I Politecni La Fe, Valencia
  - Hosp. Alvaro Cunqueiro, Vigo
- Turkey (Türkiye) (4):
  - Gazi University Medical Faculty, Ankara
  - Uludag Universitesi Tıp Fakultesi Hastanesi, Bursa
  - Ege Universitesi Tip Fakultesi, Izmir
  - Mersin University Medical Faculty, Mersin
- United Kingdom (9):
  - Fairfield General Hospital, Bury
  - Addenbrookes Hospital, Cambridge
  - Barts Health NHS Trust, London
  - Guys St Thomas Hospital, London
  - Kings College Hospital, London
  - St Georges University Hospital NHS Foundation Trust, London
  - Oxford University Hospitals NHS Foundation Trust, Oxford
  - Whiston Hospital, Prescot
  - Southampton University Hospital, Southampton

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency